CLINICAL TRIAL: NCT03757585
Title: An Open-Label Clinical Trial Conducted Via Telepsychiatry of Complementary and Alternative Treatments (Omega-3 Fatty Acids and Inositol vs. N-acetylcysteine) for the Management of Emotional Dysregulation in Youth With Non-verbal Learning Disability (NVLD) and/or Autism Spectrum Disorders (ASD)
Brief Title: Natural Treatments for the Management of Emotional Dysregulation in Youth With Non-verbal Learning Disability (NVLD) and/or Autism Spectrum Disorders (ASD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Demarest Lloyd Jr. Foundation (Unknown)
Responsible Party: Principal Investigator, Janet Wozniak, MD, Assistant Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018P002261
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Non-verbal Learning Disorder; Autism Spectrum Disorder; Autism
Keywords: autism; learning disorder; natural supplements; NAC; omega-3
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Learning Disabilities | interventions — Fatty Acids, Omega-3; Inositol; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Omega-3 Fatty Acids + Inositol (Experimental): Subjects will be treated with 1020mg QAM + 1020mg QPM of omega-3 fatty acids and inositol based on weight (subjects under 25kg: 1000mg QD; Subjects weighing 25kg or more: 2000mg QD).
  Interventions: Drug: Open-label Treatment with Omega-3 Fatty Acids + Inositol
- N-acetylcysteine (Experimental): Subjects will be treated with N-acetylcysteine capsules (subjects ages 5-12: 1800mg QD; subjects ages 13-17: 2400 mg QD) or effervescent tablets (subjects ages 5-12: 1800mg QD; subjects ages 13-17: 2700 mg QD) based on age.
  Interventions: Drug: Open-label Treatment with N-acetylcysteine

INTERVENTIONS:
Drug: Open-label Treatment with Omega-3 Fatty Acids + Inositol — Open-label Treatment with Omega-3 Fatty Acids + Inositol
  Arms: Omega-3 Fatty Acids + Inositol
Drug: Open-label Treatment with N-acetylcysteine — Open-label Treatment with acetylcysteine
  Arms: N-acetylcysteine

SUMMARY:
This study consists of a 6-week, open-label, randomized clinical trial study to compare efficacy and tolerability of the natural treatments omega-3 fatty acids, inositol, and N-acetylcysteine (NAC) in the treatment of mood dysregulation in children and adolescents with non-verbal learning disability (NVLD) or Autism Spectrum Disorder (ASD). Subjects will include youth ages 5-17 years with a non-verbal learning disability (NVLD) or autism spectrum disorder (ASD) and current symptoms of emotional dysregulation.

ELIGIBILITY:
Inclusion Criteria:

* A previous established diagnosis of non-verbal learning disability (NVLD) or DSM-V Autism Spectrum Disorder and/ or combined T-scores on the Child Behavior Checklist > 195 on the Withdrawn + Social Problems + Thought Problems subscales.
* Current symptoms of emotional dysregulation as indicated by combined T-scores on the Child Behavior Checklist > 180 on the Anxiety/Depression + Aggression + Attention subscales.
* Subjects and their caregivers must be English-speaking and have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
* Subjects and their caregivers must be willing and able to comply with all study procedures.
* Each subject and his/her authorized legal representative must understand the nature of the study. The subject's authorized legal representative must sign an informed consent document and the subject must sign an informed assent document.
* Subject must be able to swallow pills.
* Subject must have access to a computer with a camera, speaker, microphone, and internet connection.

Exclusion Criteria:

* Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
* Serious or unstable illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
* History of bleeding diathesis, including those with von Willebrand disease.
* Uncorrected hypothyroidism or hyperthyroidism.
* History of sensitivity to omega-3 fatty acids, inositol or NAC. A non-responder or history of intolerance to omega-3 fatty acid, inositol or NAC after 2 months of treatment at adequate doses as determined by the clinician.
* Severe allergies or multiple adverse drug reactions.
* Unstable or untreated seizure disorder.
* DSM-IV substance use, abuse or dependence.
* Judged clinically to be at serious suicidal risk for C-SSRS score ≥ 4.
* Current diagnosis of schizophrenia.
* Current diagnosis or symptoms of psychosis.
* IQ < 70.
* Pregnant or nursing.
* Weighs less than 12.5kg.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Wozniak, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We will use advertisements on the Internet, including advertisements posted on the Partners Clinical trials website, and flyers to recruit participants. Individuals who respond to advertising will go through a phone screen with the study coordinator or research assistant via phone and will then be screened by a study clinician.
Pre-assignment Details: Participants may also be recruited from the referral pool of existing and new patients in the Pediatric Psychopharmacology Program and the MGH Child Psychiatry Outpatient Clinic or from the pool of children screened for participation in Protocol #2019-P-000846 ("An Open-Label Clinical Trial Conducted via Telepsychiatry of Complementary and Alternative Treatments (Omega-3 Fatty Acids and Inositol vs. N-acetylcysteine) for the Management of Emotional Dysregulation in Youth").
Period: Overall Study
Arm/Group | Omega-3 Fatty Acids + Inositol | N-acetylcysteine
Started | 27 | 27
Completed | 18 | 19
Not Completed | 9 | 8

BASELINE CHARACTERISTICS:
Population: Equal numbers of baseline participants in each group.
Groups:
- Omega-3 Fatty Acid Plus Inositol: Subjects randomized to receive omega-3 fatty acids plus inositol received 2040mg (6 340mg capsules) of omega-3 fatty acids for the duration of the study. Subjects weighing 25kg or more also received 2000mg (2 1000mg capsules) of inositol per day. Children weighing less than 25kg received 1000mg (1 1000mg capsule) of inositol per day
- N-Acetylcysteine: Subjects randomized to receive NAC received NAC in either an effervescent tablet (PharmaNAC brand was chosen due to its palatability and ease of administration) or could instead opt for NAC encapsulated. For those who chose to take NAC in the effervescent tablet form, subjects age 12 and under received 1800mg daily (2 900 mg tablets) NAC and subjects age 13-17 received NAC 2700mg (3 900mg tablets) daily. For those who chose to take NAC in the capsule form, subjects age 12 and under received 1800mg (3 600mg capsules) of NAC daily and subjects age 13-17 received 2400mg (4 600mg capsules) of NAC daily.
- Total: Total of all reporting groups
Arm/Group | Omega-3 Fatty Acid Plus Inositol | N-Acetylcysteine | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 27 | 54
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 17 | 21 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 21 | 20 | 41
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 19 | 24 | 43
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Parent-Young Mania Rating Scale (P-YMRS) Score
Description: The YMRS consists of 11 items rated on a scale from 0 (symptoms not present) to 4 (symptoms extremely severe). It is used to assess manic symptoms. The YMRS score ranges from 0-60. Questions are asked about the last week. This scale is generally accepted as the main outcome measure in studies of pediatric bipolar disorder and is linked directly to the core symptoms of mania. Higher scores indicate more severe manic symptoms.
Time Frame: Baseline to 6 Weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Omega-3 Fatty Acid Plus Inositol | N-Acetylcysteine
Number analyzed (Participants) | 18 | 19
Units on a Scale | 0.0 (7.9) | -2.6 (8.1)

2. Secondary Outcome: Mean Change in the Parent-completed Children's Depression Inventory (CDI)
Description: The CDI consists of 27 items quantifying symptoms such as depressed mood, hedonic capacity, vegetative functions, self-evaluation, and interpersonal behaviors. Each item consists of three statements graded in order of increasing severity from 0 to 2; parents select the one that characterized their child's symptoms best during the past 1 week. The item scores are combined into a total depression score, which ranges from 0 to 54. A higher CDI score means a higher depressive state.
Time Frame: Baseline to 6 Weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Omega-3 Fatty Acids + Inositol | N-acetylcysteine
Number analyzed (Participants) | 18 | 19
Units on a Scale | -3.4 (7.7) | -1.3 (6.5)

3. Secondary Outcome: Mean Change in the NIMH Clinical Global Improvement Scale (CGI)
Description: The CGI-BPD-S is a clinician-rated measure of bipolar disorder severity. Severity scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The outcome reported reflects the change from baseline in CGI-BPD-S scores and negative scores represent improvement (i.e., decrease in severity from baseline).
Time Frame: Baseline to 6 Weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Omega-3 Fatty Acids + Inositol | N-acetylcysteine
Number analyzed (Participants) | 18 | 19
Units on a Scale | -1.1 (1.3) | -0.7 (1.1)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from enrollment until end of study, on average 6 weeks.
Description: Poor response to treatment, leading to drop from the study, was measured by a CGI-bipolar score that is 2 points higher (more severe) than baseline for more than 2 consecutive weeks or a P-YMRS score that is 30% higher than baseline for more than 2 consecutive weeks only if the P-YMRS is in a clinically significant range of >15. If a subject scores=d a 4 or higher on the C-SSRS, they were dropped from the study.
Arm/Group | Omega-3 Fatty Acid Plus Inositol | N-Acetylcysteine
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/27
Other Adverse Events (participants affected / at risk) | 11/27 | 13/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 Fatty Acid Plus Inositol (N=27) | N-Acetylcysteine (N=27)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 Fatty Acid Plus Inositol (N=27) | N-Acetylcysteine (N=27)
Nausea/Vomit/Diarrhea (Gastrointestinal disorders) | 6 (8) | 6 (9)
Headache (General disorders) | 3 (4) | 2 (2)
Increased Energy (General disorders) | 1 (1) | 0 (0)
Tics (Psychiatric disorders) | 1 (1) | 0 (0)
Agitated/ Irritable (Psychiatric disorders) | 0 (0) | 2 (2)
Anxious/ Worried (Psychiatric disorders) | 0 (0) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Decreased Energy (General disorders) | 0 (0) | 1 (1)
Cold/Infection/Allergy (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (3)
Dermatological (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Other (General disorders) | 3 (4) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT03757585/Prot_001.pdf
  • Statistical Analysis Plan (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT03757585/SAP_003.pdf